CLINICAL TRIAL: NCT00654654
Title: Safety and Efficacy Study of Isolagen TherapyTM in Treatment of Facial Wrinkles and Creases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT-R-007
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Facial Wrinkles and Creases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental)
  Interventions: Biological: Autologous Human Fibroblasts (azficel-T)

INTERVENTIONS:
Biological: Autologous Human Fibroblasts (azficel-T) — 1. Collection of 3 mm biopsies
  2. Two injection treatments of facial wrinkles and creases
  3. Conduct of study assessments
  Other Names: LAVIV

SUMMARY:
The purpose of this study is to evaluate the safety profile and the treatment effect of autologous human fibroblasts and placebo when administered to facial wrinkles and creases

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* High Investigator wrinkle severity assessment score
* Subject assessment of dissatisfaction of facial appearance
* Provide written informed consent and comply with the study requirements
* Negative pregnancy test at screening visit
* Healthy, non-scarred skin for biopsy

Exclusion Criteria:

* Low Investigator wrinkle severity assessment score
* Subject assessment of satisfaction of facial appearance
* Physical attributes which prevent the assessment or treatment of the facial wrinkles
* Treatment with an investigational product or procedure within 30 days or plans to participate in another clinical trial
* Previous treatment with Isolagen Therapy
* History of active autoimmune disease or organ transplantation
* Diagnosis of cancer, receiving active treatment
* History of pigmentary disorders which can affect the face
* Active or chronic skin disease
* Known genetic disorders affecting fibroblasts or collagen
* Active systemic infection
* Requires chronic antibiotic or steroidal therapy
* Use of certain cosmetic treatments & procedures
* Use of systemic agents that increase bleeding or clotting, or disorders equated with these effects
* Pregnant or lactating women or women trying to become pregnant
* Known allergic reaction to components of study treatment and/or study injection procedure
* Excessive exposure to sun or sunburn in the post-auricular area
* Subject has any disorder that may prevent compliance
* Subject who is part of the study staff, a family member or friend

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Rhonda Rand, M.D., Inc., Beverly Hills, California
  - The Laser Institute for Dermatology, Santa Monica, California
  - Winter Park and Orlando Plastic Surgery, Orlando, Florida
  - Dermatology Partners, Wellesley, Massachusetts
  - Dermatology, Laser and Vein Specialists of the Carolinas, Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 22 March 2007 and 8 August 2007
Groups:
- Autologous Fibroblasts: Patients received treatment with autologous fibroblasts to multiple facial regions
Period: Overall Study
Arm/Group | Autologous Fibroblasts
Started | 50
Completed | 43
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Fibroblasts
Number analyzed (Participants) | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 47.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  White participants | 48
  Non-white participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Subject Assessment of Wrinkles Compared to Baseline on Subject Wrinkle Assessment
Description: Subject Wrinkle Assessment was a five point ordinal scale that assessed the subject's assessment of the appearance of their face. A score of -2 (very dissatisfied) was the worst and a score of +2 (very satisfied) was the best.
Time Frame: Baseline (prior to first treatment) compared to 6 months post last treatment
Population: Number of subjects for whom data were available from the assessment visit, 6 months after the final treatment
Measure: Number; unit: participants
Groups:
- Autologous Fibroblasts: Patients treated with autologous human fibroblasts
Arm/Group | Autologous Fibroblasts
Number analyzed (Participants) | 41
participants
  Change = -1 (worse) | 2
  Change = 0 (no change) | 5
  Change = +1 (better) | 15
  Change = +2 (better) | 11
  Change = +3 (better) | 7
  Change = +4 (better) | 1

2. Primary Outcome: Independent Panel Global Improvement Assessment Compared to Baseline
Description: An independent panel of physicians reviewed photographs of subjects at baseline and 6 months after final study treatment and provided a score for improvement in appearance on the Global Improvement Assessment. The Global Improvement Assessment was a four point ordinal scale with 0 (No improvement) as the worst score and 3 (Marked Improvement) the best.
Time Frame: Baseline (prior to treatment) compared to 6 months post last treatment
Population: Number of patients for whom data were available
Measure: Number; unit: participants
Arm/Group | Autologous Fibroblasts
Number analyzed (Participants) | 44
participants
  No improvement | 10
  Mild improvement | 29
  Moderate improvement | 5
  Marked improvement | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for six months after final study treatment
Groups:
- Active: Patients treated with autologous human fibroblasts
Arm/Group | Active
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=50)
Dehydration (Metabolism and nutrition disorders) | 1 (1) — SAE occurred prior to study treatment
Alcoholism (Psychiatric disorders) | 1 (1) — SAE occurred prior to study treatment
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — SAE occurred after study treatment, and was considered unrelated by the Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=50)
Acne (Skin and subcutaneous tissue disorders) | 4
Headache (Nervous system disorders) | 3
Injection site bruising (General disorders) | 5
Injection site erythema (General disorders) | 6
Injection site nodule (General disorders) | 4
Injection site pain (General disorders) | 3
Injection site swelling (General disorders) | 5
Nasophayngitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications or presentations by the Investigator or his associates, were required to be submitted to the sponsor for review and approval prior to publication or presentation in any form.